CLINICAL TRIAL: NCT05900219
Title: A Single-arm, Open, Multicenter Phase II Study to Evaluate the Efficacy and Safety of HL-085 Capsules Combined With Vemurafenib in the Treatment of BRAF V600E Mutated Patients With Unresectable Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC)
Brief Title: Efficacy and Safety of HL-085 Combined With Vemurafenib in BRAF V600E Patients With Non-small Cell Lung Cancer: a Phase II Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Kechow Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL-085-203
Record Dates: First submitted 2023-05-29; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Non-small-cell Lung Cancer
Keywords: BRAF V600E mutation; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental): The treatment regimen was HL-085 9mg BID+ Vemurafenib 720mg BID oral administration
  Interventions: Drug: HL-085+Vemurafenib

INTERVENTIONS:
Drug: HL-085+Vemurafenib — The treatment regimen was HL-085 9mg BID+ Vemurafenib 720mg BID oral administration for 21 days per cycle. The primary efficacy endpoint in this study was the ORR assessed by the Independent Review Committee (IRC) according to the RECIST 1.1

SUMMARY:
This is a single-arm, open, multicenter phase II clinical study to evaluate the efficacy and safety of HL-085 capsules combined with Vemurafenib in the treatment of BRAF V600E mutated patients with unresectable locally advanced or metastatic NSCLC. Meanwhile, to explore the relationship between pop-PK characteristics, efficacy and safety in the treatment of HL-085 combined with Vemurafenib

DETAILED DESCRIPTION:
This study was intended to be divided into two study cocohorts. Cohort one was BRAF V600E mutated NSCLC patients who had not received systemic treatment (first-line). Cohort 2 included patients with BRAF V600E mutated NSCLC who had received systemic therapy (second-line and above); There were 30 patients in cohort 1 and 39 in cohort 2, a total of 69 evaluable cases. A sample size of 73 patients with advanced NSCLC with BRAF V600E mutation (32 /41, respectively) was calculated at a 5% shedding rate. All patients in the first/second line and above were eligible for inclusion. The treatment regimen was HL-085 9mg BID+ Vemurafenib 720mg BID oral administration for 21 days per cycle. The primary efficacy endpoint in this study was the ORR assessed by the Independent Review Committee (IRC) according to the RECIST 1.1 Efficacy Evaluation Criteria for solid tumors. Subjects were evaluated for tumor imaging every 6 weeks (±7 days), and for complete response (CR) or partial response (PR) at the first imaging assessment, reconfirmation was performed at ≥4 weeks. Safety will be assessed by vital signs, physical examination, ECOG score, clinical laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, myocardial enzymes), 12-lead electrocardiogram (ECG), echocardiogram (ECHO) examination, and incidence and severity of AE.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Male or female aged 18-75 (inclusive) at the time of signing the informed consent;
  2. Patients with locally advanced or metastatic stage IIIb, IIIc, or IV NSCLC (according to the AJCC Eighth Edition TNM staging system for lung cancer) who are confirmed by histopathology/cytology and cannot be resected by surgery can be included in the group without or after systemic treatment;
  3. At baseline, genetic testing reports of BRAF V600E mutation can be provided;
  4. The time interval between the end of the last anti-tumor therapy and the first administration of the study drug meets the following requirements: ≥4 weeks for cytotoxic drugs and cellular immunotherapy; PD-1/PD-L1/CTLA-4≥6 weeks; Small-molecule targeted drugs ≥2 weeks or 5 half-lives of drugs (whichever is longer); Mitomycin/nitrosourea ≥6 weeks; End time of radiotherapy ≥4 weeks (palliative local radiotherapy for pain relief ≥2 weeks), radiotherapy related adverse reactions recovered;
  5. ECOG PS score 0-1;
  6. Expected survival > 3 months;
  7. At least one measurable lesion in line with the RECIST v1.1 definition at baseline (if the lesion at the site of previous radiotherapy is selected as the target lesion, this lesion has obvious evidence of progression);
  8. The level of organ function and related laboratory indicators must meet the following requirements:

     * Neutrophil count absolute value (ANC) ≥ 1.5×109/L; Platelet count ≥ 100×109/L; Hemoglobin ≥ 90g/L;
     * Blood biochemistry: serum total bilirubin ≤1.5 times the upper limit of normal value (ULN); For Gilbert syndrome patients, TBIL≤3×ULN; AST/ALT≤3 ULN (Allow AST/ALT≤5 ULN when liver metastasis occurs); Serum creatinine ≤1.5 ULN; Albumin ≥30 g/L;
     * Coagulation: prothrombin time (PT) ≤ 1.5x ULN or activated partial thrombin time (APTT) ≤ 1.5x ULN;
     * Creatine phosphokinase (CPK) and (hypersensitive) troponin (cTnI/T) are within normal ranges;
  9. The serum pregnancy test results of fertile women must be negative within 7 days prior to the first dosing, and female subjects are willing to use adequate contraception during the trial and for at least 6 months after the last dosing of the study drug. Male subjects must consent to use contraception (non-drug or tool contraception) for at least 6 months from the start of the study until the final dose;
  10. The subjects voluntarily participated in the study and signed the informed consent. The subjects had good compliance and could cooperate with the follow-up.

Exclusion Criteria:

* Exclusion Criteria:

  1. Patients who are known to have an allergic reaction to any BRAF and/or MEK inhibitors and their excipients or have an allergic predisposition;
  2. Patients with EGFR mutation, ALK fusion and other positive driver genes;
  3. Previous history of antitumor and surgical treatment conforms to any of the following:

     * Being in the treatment phase of another clinical study within 4 weeks prior to initial dosing (except for patients participating in overall survival follow-up);
     * Has undergone major surgery or has not fully recovered from previous invasive procedures within 4 weeks prior to initial dosing (other than baseline tumor biopsy);
     * Previous use of MEK inhibitors, including but not limited to trametinib, smeitinib, caubitinib, pimetinib, and/or BRAF inhibitors, including but not limited to vermofinib, dalafenib, and Conefenib;
  4. Symptomatic or untreated brain metastases, meninges, or spinal cord compression (imaging instability, symptomatic lesion, need for hormonal or dehydration treatment); Subjects with asymptomatic and stable brain metastases (brain lesions ≥4 weeks stable without progression) could be enrolled;
  5. Pleural effusion, pericardial effusion and abdominal effusion that still cannot be controlled after clinical intervention;
  6. Patients with malignancies other than the type of tumor studied within 3 years prior to initial administration, except local cancers that have been apparently cured or have been free of disease for at least 3 years, such as basal or squamous cell skin cancer, superficial bladder cancer, prostate cancer in situ, cervical cancer in situ, or ductal carcinoma in situ of the breast;
  7. Patients who have previously received allogeneic bone marrow transplantation or organ transplantation;
  8. Previous or current retinal diseases, such as retinal venous obstruction (RVO), retinal arterial obstruction (RAO), retinal vasculitis, diabetic retinopathy, hypertensive retinopathy, retinal telangiectasis (Costs disease), retinal pigment epithelium detachment (RPED), etc.;
  9. Patients with past or current interstitial lung disease, including clinically significant radiation pneumonia (i.e. affecting activities of daily living or requiring intervention);
  10. Past or current neuromuscular diseases associated with elevated CPK (e.g., inflammatory myopathy, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy, rhabdomyolysis syndrome);
  11. Bleeding symptoms ≥ Grade 3 as defined in NCI CTCAE v5.0 occurred within 4 weeks prior to initial administration;
  12. Subjects with impaired heart function or clinically significant cardiovascular and cerebrovascular diseases, including any of the following:

      * Acute myocardial infarction, unstable angina, or acute cerebral infarction
      * Stent implantation during coronary angioplasty or within 6 months prior to initial administration
      * Clinically significant unstable arrhythmias (atrial fibrillation, etc.)
      * Congestive heart failure of grade II or higher as defined by New York Heart Society (NYHA) standards; Note: Subjects with grade 1 abnormal heart valve morphology recorded by ECHO (≥ Grade 2) were admitted, but subjects with moderate valve thickening were excluded;
      * QT interval (QTcF) ≥ 480 msec corrected using the Fridericia formula;
      * Left ventricular ejection fraction (LVEF) < 55%;
      * Implantable defibrillators;
      * Refractory hypertension (at least 3 consecutive months of use of at least 3 antihypertensive drugs, still unable to control blood pressure within the normal range);
  13. Inability to swallow capsules or refractory nausea and vomiting, malabsorption, extracorporeal bile shunt, or any significant small intestine resection that might prevent full absorption of the study drug; Chronic atrophic gastritis and gastroduodenal ulcer with bleeding risk;
  14. Human immunodeficiency virus (HIV) antibody positive, syphilis antibody (Anti-TP) positive, hepatitis C virus (HCV) antibody positive and HCV-RNA positive, hepatitis B virus surface antigen (HBsAg) positive and HBV-DNA positive (HBsAg positive requires further HBV DNA testing, HBV DNA≥200 IU/ml, or ≥103 copy number /ml);
  15. Strong inducers that affect cytochrome P450 (CYP) isoenzymes (CYP2C9, CYP3A4) that are prohibited by protocol, strong inhibitors or drugs with a narrow therapeutic window through CYP1A2 metabolism should continue to be used within 7 days prior to initial administration or during the study period;
  16. There was > grade 1 unmitigated toxicity associated with prior antitumor therapy prior to initial administration. Alopecia, skin pigmentation, grade 2 neurotoxicity due to prior platinum therapy, asymptomatic hypothyroidism due to immune checkpoint inhibitors requiring hormone replacement therapy, and medicated hyperglycemia were excluded;
  17. The presence of any serious and/or unstable pre-existing condition, mental illness, or other condition that may interfere with the subject's safety, obtaining informed consent, or complying with study procedures. Including, but not limited to, severe diabetes (fasting blood glucose ≥13.9mmol/L), active infections (such as active tuberculosis), active bleeding, or other serious diseases requiring systematic treatment;
  18. lactating women;
  19. The investigator determined that the subjects had a serious or uncontrolled systemic disease that would make them unfit to participate in the study or would affect protocol compliance or significantly interfere with the correct assessment of the safety, toxicity, or efficacy of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-24 (Estimated); Primary Completion 2025-09-24 (Estimated); Study Completion 2025-09-24 (Estimated)

PRIMARY OUTCOMES:
ORR | through study completion, an average of 1 year
  Defined as the proportion of subjects with an optimal response of CR or PR over the course of the study from enrollment to disease progression (PD), dominated by IRC assessment. CR and PR must be reassessed for confirmation ≥4 weeks after first meeting mitigation criteria;

SECONDARY OUTCOMES:
DOR | through study completion, an average of 1 year
  Defined as the time from the first CR or PR evaluation of tumor efficacy to the first occurrence of PD or death from any cause (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, phD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science

IPD SHARING:
Plan to Share IPD: No